CLINICAL TRIAL: NCT02139800
Title: Sustained Aeration of Infant Lungs Trial
Acronym: SAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 819208; 1U01HD072906-01A1 (NIH)
Record Dates: First submitted 2014-05-08; First posted 2014-05-15 (Estimated); Results first posted 2020-06-25 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Preterm Birth; Extreme Prematurity
Keywords: Neonatal resuscitation; Extreme Low Gestational Age Newborn (ELGAN); Delivery Room; Continuous positive airway pressure (CPAP); Positive pressure ventilation (PPV); Sustained inflation
MeSH Terms: conditions — Premature Birth | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm-Standard of care (Active Comparator): Control Arm-Respiratory support using Standard of Care positive-end expiratory pressure/continuous positive airway pressure (PEEP/CPAP) of 5-7 cm H2O compared to Sustained Inflation intervention
  Interventions: Procedure: Standard of Care
- Sustained Intervention (Experimental): Administer delivery room respiratory support using a Sustained Inflation (SI) intervention and expiratory pressure/continuous positive airway pressure (PEEP/CPAP) of 5-7 cm H2O
  Interventions: Procedure: Sustained Inflation

INTERVENTIONS:
Procedure: Sustained Inflation — The first sustained inflation will use inflation pressure of 20 cm H20 for 15 seconds
  Arms: Sustained Intervention
Procedure: Standard of Care — Newborn Resuscitation Program (NRP) Guidelines using a standard PEEP/CPAP of 5-7 cm H2O as compared to the Sustained Inflation intervention
  Arms: Control Arm-Standard of care

SUMMARY:
This study is a 2-arm randomized, controlled, multi-center clinical trial to determine which of two strategies at birth are best to optimally aerate the lung of preterm infants. Specifically we will determine in 600 infants of 23-26 weeks gestational age (GA) requiring respiratory support at birth which of two lung opening strategies - either a standard PEEP/CPAP of 5-7 cm H2O in the delivery room (DR), as compared to early lung recruitment using Sustained Inflation (SI) in the DR, will result in a lower rate of the combined endpoint of death or bronchopulmonary dysplasia (BPD) at 36 weeks gestational age.

Hypotheses:

1. Early lung recruitment with SI superimposed upon standard PEEP/CPAP in the DR will reduce the need for mechanical ventilation in the first seven days of life, and reduce need for surfactant use; and
2. A policy of DR SI on standard PEEP/CPAP recruitment will confer better outcomes at 36 weeks post-menstrual age (PMA) than standard PEEP/CPAP

DETAILED DESCRIPTION:
The SAIL trial aims to provide evidence for changing policy or standard of care. The context of this trial is an unacceptable rate of poor long-term outcomes of preterm infants born as Extremely Low Gestational Age Newborns (ELGAN) <1000 g birthweight (BW), but especially for those born between 23-26 weeks' gestational age (GA). Such infants are the most vulnerable and immature in all organ systems, including the lungs and the brain. These infants are at high risk of death and bronchopulmonary dysplasia (BPD) during their initial hospitalization, neurodevelopmental impairment (NDI) and pulmonary problems in infancy and childhood.

The SAIL trial focuses on facilitating the difficult transition of these most vulnerable infants from a liquid filled in-utero lung to an ex-utero air-filled lung. Sustained Inflation (SI) is a promising delivery room (DR) intervention, with evidence of short-term efficacy with minimal risk of additional harm beyond current standard accepted Newborn Resuscitation Program (NRP) Guidelines. This protocol proposes a fully informed consenting procedure. We propose to evaluate the impact of a SI in the DR on the need for mechanical ventilation in the first week of life which would also impact mortality rates and the incidence and severity of BPD.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) at least 23 weeks but less than 27 completed weeks by best obstetrical estimate
* Requiring resuscitation/respiratory intervention at birth -"apneic, labored breathing, gasping" (as defined in NRP 2011 AAP 6th Edition p.45)

Exclusion Criteria:

* Considered non-viable by the attending neonatologist
* Refusal of antenatal informed consent
* Known major anomalies, pulmonary hypoplasia
* Mothers who are unable to consent for their medical care and who do not have a surrogate guardian will not be approached for consent

Ages: 23 Weeks to 26 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 460 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haresh Kirpalani, BM, MSc, Principal Investigator — Children's Hospital of Philadelphia; Peter Davis, MD, FRAXP, Principal Investigator — Royal Women's Hospital, Melbourne, Australia; Helmut Hummler, MD, Principal Investigator — Children's Hospital, University of Ulm, Ulm Germany; Martin Keszler, MD, Principal Investigator — Women & Infants Hospital of Rhode Island, Providence, RI; GianLuca Lista, MD, Principal Investigator — Ospedale dei Bambini, Milan Italy; Arjan te_Pas, MD, Principal Investigator — Leiden University Medical Center, Leiden, Netherlands
Locations (21):
- United States (9):
  - Loma Linda University, Loma Linda, California
  - University of California, Davis Children's Hospital, Sacramento, California
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - Christiana Care, Newark, Delaware
  - University of Michigan, Ann Arbor, Michigan
  - Wake Med Health, Raleigh, North Carolina
  - Hospital of the Univerity of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
- Australia (2):
  - Mater Mother's Hospital, Brisbane, Queensland
  - Royal Women's Hospital, Melbourne
- Academic Teaching Hospital, Landeskrankenhaus Feldkirch, Feldkirch, Austria
- Royal Alexandra Hospital,, Edmonton, Canada
- Germany (2):
  - University of Freiburg, Freiburg im Breisgau
  - Children's Hospital, University of Ulm, Ulm
- Ospedale dei Bambini, Milan, Italy
- Netherlands (2):
  - Emma Children's Hospital, AMC, Amsterdam
  - Leiden University Medical Center, Leiden
- KK Women's and Children's Hospital, Singapore, Singapore
- South Korea (2):
  - Seoul National University Children's Hospit, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Owen LS, Foglia EE, Ratcliffe SJ, Simma B, Katheria AC, Te Pas A, Onland W, van Kaam AH, Keszler M, Kirpalani H, Davis PG. Alternative consent processes in a neonatal resuscitation trial (SAIL): secondary analysis of an open-label, international, multicentre, randomised trial. Lancet Child Adolesc Health. 2025 Oct;9(10):698-706. doi: 10.1016/S2352-4642(25)00185-3. Epub 2025 Aug 12. PMID 40816312
- [Derived] Foglia EE, Kirpalani H, Ratcliffe SJ, Davis PG, Thio M, Hummler H, Lista G, Cavigioli F, Schmolzer GM, Keszler M, Te Pas AB. Sustained Inflation Versus Intermittent Positive Pressure Ventilation for Preterm Infants at Birth: Respiratory Function and Vital Sign Measurements. J Pediatr. 2021 Dec;239:150-154.e1. doi: 10.1016/j.jpeds.2021.08.038. Epub 2021 Aug 25. PMID 34453917
- [Derived] Kirpalani H, Keszler M, Foglia EE, Davis P, Ratcliffe S. Considering the Validity of the SAIL Trial-A Navel Gazers Guide to the SAIL Trial. Front Pediatr. 2019 Nov 27;7:495. doi: 10.3389/fped.2019.00495. eCollection 2019. PMID 31828052
- [Derived] Kirpalani H, Ratcliffe SJ, Keszler M, Davis PG, Foglia EE, Te Pas A, Fernando M, Chaudhary A, Localio R, van Kaam AH, Onland W, Owen LS, Schmolzer GM, Katheria A, Hummler H, Lista G, Abbasi S, Klotz D, Simma B, Nadkarni V, Poulain FR, Donn SM, Kim HS, Park WS, Cadet C, Kong JY, Smith A, Guillen U, Liley HG, Hopper AO, Tamura M; SAIL Site Investigators. Effect of Sustained Inflations vs Intermittent Positive Pressure Ventilation on Bronchopulmonary Dysplasia or Death Among Extremely Preterm Infants: The SAIL Randomized Clinical Trial. JAMA. 2019 Mar 26;321(12):1165-1175. doi: 10.1001/jama.2019.1660. PMID 30912836
- [Derived] Foglia EE, Te Pas AB. Sustained Lung Inflation: Physiology and Practice. Clin Perinatol. 2016 Dec;43(4):633-646. doi: 10.1016/j.clp.2016.07.002. PMID 27837749
- [Derived] Foglia EE, Owen LS, Thio M, Ratcliffe SJ, Lista G, Te Pas A, Hummler H, Nadkarni V, Ades A, Posencheg M, Keszler M, Davis P, Kirpalani H. Sustained Aeration of Infant Lungs (SAIL) trial: study protocol for a randomized controlled trial. Trials. 2015 Mar 15;16:95. doi: 10.1186/s13063-015-0601-9. PMID 25872563

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Arm-Standard of Care | Sustained Intervention
Started | 224 | 236
Completed (These infants have completed their 36 week PMA primary outcome) | 211 | 215
Not Completed | 13 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm-Standard of Care | Sustained Intervention | Total
Number analyzed (Participants) | 211 | 215 | 426
Age, Customized [Count of Participants; unit: Participants] — Infants were included in the study based on their gestational age. - include GA strata
  Participants
    23-24 weeks GA | 75 | 76 | 151
    25-26 weeks GA | 136 | 139 | 275
Sex: Female, Male [Count of Participants; unit: Participants] — The sex of the infants are included below.
  Participants
    Female | 108 | 96 | 204
    Male | 103 | 119 | 222
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Maternal race/ethnicity is listed below
  Participants
    White | 110 | 148 | 258
    Black | 50 | 29 | 79
    Asian | 23 | 18 | 41
    Other | 28 | 20 | 48
Region of Enrollment [Number; unit: participants]
  Canada | 23 | 20 | 43
  Netherlands | 50 | 56 | 106
  Austria | 6 | 5 | 11
  South Korea | 5 | 3 | 8
  Singapore | 0 | 1 | 1
  United States | 61 | 66 | 127
  Italy | 11 | 13 | 24
  Australia | 35 | 30 | 65
  Germany | 20 | 21 | 41
Consent Type [Number; unit: participants]
  Antenatal | 113 | 122 | 235
  Deferred | 98 | 93 | 191
Maternal Age [Median (Inter-Quartile Range); unit: years] | 30.5 [26.0 to 34.9] | 31.1 [26.5 to 35.4] | 30.9 [26.3 to 35.2]

OUTCOME MEASURES:

1. Primary Outcome: Combined Outcome of Death or Bronchopulmonary Dysplasia
Description: To determine in infants born at 23-26 weeks gestational age requiring respiratory support at birth, which of two treatment strategies when compared, results in a lower rate of the combined endpoint of death or bronchopulmonary dysplasia.
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm-Standard of Care | Sustained Intervention
Number analyzed (Participants) | 211 | 215
Participants | 125 | 137

2. Secondary Outcome: Oxygen Profile Over First 24 Hours
Description: Oxygen profile over first 24 hours post delivery room using hourly FiO2 records
Time Frame: First 24 hours post delivery
Reporting Status: Not Posted

3. Secondary Outcome: Oxygen Profile With Highest FiO2 Level up to 48 Hours
Description: Highest FiO2 level recorded during the first 48 hours post DR
Time Frame: 48 hours of life
Reporting Status: Not Posted

4. Secondary Outcome: Heart Rate in the Delivery Room (DR)
Description: Categorical variable with 3 levels: <60, 60-100, >100
Time Frame: First 30 seconds of life in DR
Reporting Status: Not Posted

5. Secondary Outcome: Detailed Status on Departure From the Delivery Room (DR)
Description: Type of respiratory support (CPAP, PPV) and Fraction of Inspired Oxygen (FiO2) on departure from DR
Time Frame: Resuscitation time will vary - 1 to 30 minutes
Reporting Status: Not Posted

6. Secondary Outcome: Use of Inotropes on Arrival in NICU
Description: Circulatory support post-delivery room
Time Frame: First 48 hours of life
Reporting Status: Not Posted

7. Secondary Outcome: Need for Intubation in Delivery Room
Description: Need for intubation in delivery room during the first 30 seconds to 24 hours of age
Time Frame: First 30 seconds to 24 hours of life
Reporting Status: Not Posted

8. Secondary Outcome: Pressure-volume Characteristics in the Delivery Room (DR)
Description: Pressure-volume characteristics in the Delivery room (DR) expected within 30 minutes
Time Frame: Expected average 30 minutes
Reporting Status: Not Posted

9. Secondary Outcome: Pneumothorax or New Chest Drains in the First 48 Hours of Life
Description: Chest x-ray reports showing pneumothorax or new chest drains in the first 48 hours of life
Time Frame: First 48 hours of life
Reporting Status: Not Posted

10. Secondary Outcome: Duration of Any Chest Drain In-situ Post-DR
Description: Duration of any chest drain in-situ post-DR during hospitalization - up to 36 weeks Post Menstrual Age (PMA)
Time Frame: During hospitalization - up to 36 weeks Post Menstrual Age (PMA)
Reporting Status: Not Posted

11. Secondary Outcome: Intraventricular Hemorrhage by All Grades
Description: Head ultrasound and/or MRI findings of intraventricular hemorrhage by all grades focusing on grades 3 and 4 by 48 hour and by day 10
Time Frame: 48 hours to 10 days
Reporting Status: Not Posted

12. Secondary Outcome: Chest X-ray Between Days 7-10
Description: Chest x-ray between the first 7-10 days of life
Time Frame: First 7-10 days of life
Reporting Status: Not Posted

13. Secondary Outcome: Death or Need for Positive Pressure Ventilation
Description: Death or need for positive pressure ventilation during the first 7 days of life
Time Frame: First 7 days of life
Reporting Status: Not Posted

14. Secondary Outcome: Highest FiO2 and Area Under the FiO2 Curve for the First Week of Life
Description: Highest FiO2 and Area under the FiO2 curve during the first 7 days of life
Time Frame: First 7 days of life
Reporting Status: Not Posted

15. Secondary Outcome: Pneumothorax and Pulmonary Interstitial Emphysema (PIE)
Description: Pneumothorax and pulmonary interstitial emphysema (PIE) during the first 10 days of life
Time Frame: First 10 days of life
Reporting Status: Not Posted

16. Secondary Outcome: Survival to Discharge Home Without BPD, Retinopathy of Prematurity (Grades 3 & 4), or Significant Brain Abnormalities on Head Ultrasound
Description: Survival to discharge home without BPD, retinopathy of prematurity (grades 3 & 4), or significant brain abnormalities on head ultrasound with an expected discharge between 36-40 weeks PMA
Time Frame: Expected discharge between 36 - 40 weeks PMA
Reporting Status: Not Posted

17. Secondary Outcome: Duration of Respiratory Support (Ventilation, CPAP, Supplemental Oxygen)
Description: Duration of respiratory support (ventilation, CPAP, supplemental oxygen) during hospitalization upto 36 weeks Post Menstrual Age (PMA)
Time Frame: During hospitalization - up to 36 weeks Post Menstrual Age (PMA)
Reporting Status: Not Posted

18. Secondary Outcome: Death in Hospital
Description: Death in hospital during expected hospitalization of 23-40 weeks PMA
Time Frame: During expected hospitalization 23 - 40 weeks PMA
Reporting Status: Not Posted

19. Secondary Outcome: Retinopathy of Prematurity (ROP) Stage 3 or Greater Requiring Treatment
Description: Retinopathy of prematurity (ROP) stage 3 or greater requiring treatment at 36 weeks
Time Frame: 36 weeks
Reporting Status: Not Posted

20. Secondary Outcome: Use of Postnatal Steroids for Treatment of BPD
Description: Use of postnatal steroids for treatment of BPD during hospitalization up to 36 weeks Post Menstrual Age (PMA)
Time Frame: During hospitalization - up to 36 weeks Post Menstrual Age (PMA)
Reporting Status: Not Posted

21. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay with average discharge between 36-40 weeks PMA
Time Frame: Average discharge between 36 - 40 weeks PMA
Reporting Status: Not Posted

22. Secondary Outcome: Neurodevelopmental and Respiratory Outcome at 22-26 Months Corrected Gestational Age
Description: Neurodevelopmental and respiratory outcome at 22-26 months corrected gestational age
Time Frame: 22-26 months corrected gestational age
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from birth to discharge, death or 44 weeks PMA whichever occurred first
Arm/Group | Control Arm-Standard of Care | Sustained Intervention
All-Cause Mortality (participants affected / at risk) | 35/211 | 48/215
Serious Adverse Events (participants affected / at risk) | 51/211 | 45/215
Other Adverse Events (participants affected / at risk) | 146/211 | 157/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm-Standard of Care (N=211) | Sustained Intervention (N=215)
Death (Pregnancy, puerperium and perinatal conditions) | 3 | 16 — Within the first 48 hours post delivery
Administration of epinephrine or chest compressions (Surgical and medical procedures) | 8 | 6 — Within the first 48 hours post delivery
Pneumothorax (Pregnancy, puerperium and perinatal conditions) | 19 | 11 — Within the first 10 days of life
Pulmonary Interstitial Emphysemia (PIE) (Respiratory, thoracic and mediastinal disorders) | 6 | 7 — Within the first 10 days of life
Grade 3 or 4 IVH (Pregnancy, puerperium and perinatal conditions) | 22 | 21 — Within the first 10 days of life
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm-Standard of Care (N=211) | Sustained Intervention (N=215)
FiO2>=0.4 for >=2 hrs in first 2 DOL (Surgical and medical procedures) | 52 | 50
IVH Grade 1/2 within first 10 days of life (Pregnancy, puerperium and perinatal conditions) | 44 | 51
>30% oxygen at 28 days of life (Surgical and medical procedures) | 76 | 66
Mechanical support at 28 days of life (Surgical and medical procedures) | 91 | 84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT02139800/Prot_000.pdf
  • Statistical Analysis Plan (2014-04-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT02139800/SAP_001.pdf